CLINICAL TRIAL: NCT06389201
Title: Pretreatment With HCQ Before Radiotherapy and Chemotherapy in Advanced NPC Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024HCQ
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: autophagy; tumor dormancy; nasopharyngeal carcinoma; recurrence; metastasis
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Recurrence; Neoplasm Metastasis | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pretreatment with an autophagy inhibitor (HCQ) before chemotherapy and radiotherapy (Experimental): Hydroxychloroquine (HCQ), is used one day before chemotherapy and radiotherapy, 400-600mg, oral tablet, once. During chemotherapy and radiotherapy, HCQ maintenance dose is 200-400mg daily.
  Interventions: Drug: HCQ
- Receive placebo before and during chemotherapy and radiotherapy (Placebo Comparator): Placebos are used one day before chemotherapy and radiotherapy, and during the therapy.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: HCQ — HCQ, 400-600mg, oral tablet, once, one day before chemotherapy and radiotherapy. During therapy, HCQ maintenance dose is 200-400mg daily.
  Other Names: Hydroxychloroquine
  Arms: Pretreatment with an autophagy inhibitor (HCQ) before chemotherapy and radiotherapy
Other: Placebo — Placebo, oral tablet, once, one day before chemotherapy and radiotherapy. During therapy, placebo maintenance oral tablet once daily.
  Arms: Receive placebo before and during chemotherapy and radiotherapy

SUMMARY:
Dormant cancer cells that survive anti-cancer therapy can lead to cancer recurrence and disseminated metastases that prove fatal in most cases. Recently, specific dormant polyploid giant cancer cells (PGCC) have drawn the investigators' attention because of their association with the clinical risk of nasopharyngeal carcinoma (NPC) recurrence, as demonstrated by previous clinical data. In study, the investigators report the biological properties of PGCC, and reveal that autophagy is a critical mechanism of PGCC induction. Moreover, pharmacological inhibition of autophagy greatly impaired PGCC formation, significantly suppressing metastasis and improving survival in a mouse model. Mechanistically, chemotherapeutic drugs partly damaged mitochondria, and activated autophagy to promote PGCC formation. High numbers of PGCCs correlated with shorter recurrence time and worse survival outcomes in NPC patients. Collectively, these findings suggest a therapeutic approach of targeting dormant PGCCs in cancer.

Pretreatment with an autophagy inhibitor (HCQ) before chemotherapy and radiotherapy could prevent formation of therapy-induced dormant polyploid giant cancer cells, thereby reducing recurrence and metastasis of nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Although the majority of patients with nasopharyngeal carcinoma (NPC) do not present with overt metastases at diagnosis, a significant number succumb to disseminated disease years after the successful treatment of the primary tumor. Thus, late NPC recurrence may be the result of rare and elusive dormant cancer cells hiding in specialized niches being reactivated by specific signals. The concept of cancer dormancy has been described for the most common solid and hematological cancers; however, the dormant cancer cells in NPC remain largely uncharacterized.

Although many factors contribute toward cancer cell dormancy, recent studies have demonstrated that cancer therapy can induce cellular dormancy. Indeed, therapy-induced dormancy has been shown to lead to durable proliferation arrest, resulting in the formation of polyploid giant cancer cells (PGCCs), which are a unique sub-population of cancer cells that contribute toward the heterogeneity of solid tumors. Unlike regular-sized diploid cancer cells, PGCCs display distinct morphological features, including a large cytoplasmic area and a high genomic content contained within a single highly enlarged nucleus or multiple nuclei. Despite being present in low numbers, the frequency of PGCCs increases markedly after exposure to hypoxia and therapeutic interventions such as radiotherapy and chemotherapies.

The investigators' findings, which used a highly relevant clinical orthotopic model of imageable NPC and clinical data, suggest that autophagy inhibition (HCQ) prevents therapy-induced dormant PGCC formation and thereby prevents NPC metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of NPC.
* Have not received any cancer therapies
* Must provide informed consent

Exclusion Criteria:

* With metastasis before the first treatment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2034-08-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence and metastasis | Five to Ten years.
  After the patients are diagnosed and treated, CT scans is used semi-annually to determine the progression, recurrence and metastasis of tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Bo You, Doctor, Principal Investigator — Department of Otorhinolaryngology-Head and Neck Surgery, Affiliated Hospital of Nantong University
Locations (1):
- Bo You, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan, informed consent form, clinical study report, and analytic code will be shared to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Two years after this clinical trial finished.
Access Criteria: Researchers must clearly state the purpose of their study and ensure it aligns with the scientific objectives of the data sharing initiative. A detailed research plan, including research design, data analysis methods, and expected results, should be provided to ensure the data is used in a reasonable and effective manner. Additionally, researchers must outline data security and privacy protection measures to ensure the safe storage, transmission, and use of the data in compliance with relevant regulations and policies.